CLINICAL TRIAL: NCT04686773
Title: Open-label, Non-randomized, Non-comparative, Phase II Study in Adult Subjects to Assess Safety and Immunogenicity of Combination of AZD1222, a Non-replicating ChAdOx1 Vector Vaccine, and rAd26-S, a Recombinant Adenovirus Type 26 Component of Gam-COVID-Vac Vaccine, for COVID-19 Prevention
Brief Title: Open-label, Non-randomized, Non-comparative, Phase II Study of Safety and Immunogenicity of Combination of AZD1222 and rAd26-S for COVID-19 Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: AstraZeneca (Industry); Russian Direct Investment Fund (Industry); The Gamaleya National Center of Epidemiology & Microbiology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CV03872092
Record Dates: First submitted 2020-12-25; First posted 2020-12-29 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Severe acute respiratory syndrome coronavirus 2; 2019-nCoV; 2019 novel coronavirus; Respiratory disease; lung disease; COVID-19; coronavirus
MeSH Terms: conditions — COVID-19; Respiration Disorders; Lung Diseases; Coronavirus Infections | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD1222 5×10^10 vp + rAd26-S (1.0±0.5) х 10^11vp (Experimental): Subjects will receive 1 intramuscular (IM) injection of 5×10^10 viral particles (nominal) of AZD1222 on Day 1 followed by rAd26-S 1×10^11 viral particles (nominal) on Day 29 of the study.
  Interventions: Biological: AZD1222; Biological: rAd26-S

INTERVENTIONS:
Biological: AZD1222 — AZD1222 (0.5 ml per dose) contains:
  Active substance: ChAdOx1 nCoV-19, a replicant-deficient simian adenoviral vector in the amount of 5 х 10^10 particles per dose.
  Solution for intramuscular injection, supplied in vials (5 mL, up to 10 doses per vial) in a carton box.
  Other Names: AZ_VACCINE_COVID-19; (previously called ChAdOx1 nCoV-19)
Biological: rAd26-S — Component I (0.5 ml per dose) contains:
  Active substance: recombinant adenovirus serotype 26 particles containing the SARS-CoV-2 protein S gene, in the amount of (1.0±0.5) х 10^11 particles per dose.
  Solution for intramuscular injection, supplied in vials (3 mL, 5 doses per vial) in a carton box
  Other Names: Gam-COVID-Vac combined vector vaccine (Component I)

SUMMARY:
The purpose of the study is to assess safety and immunogenicity of heterologous booster vaccine containing combination of AZD1222 and rAd26-S (one of components of Gam-COVID-Vac vaccine) in adult subjects aged ≥ 18 years old to prevent COVID-19 spread.

DETAILED DESCRIPTION:
This clinical study is a prospective, single-center, open-label, non-comparative, non-randomized single-arm study. It will enroll adult subjects aged ≥ 18 years old with absence of active COVID-19 infection to be verified by the results of reverse transcription polymerase chain reaction (RT-PCR).

100 subjects meeting inclusion criteria are expected to be screened, 100 of them meeting eligibility criteria will receive one intramuscular injection of AZD1222 vaccine at 5×10^10 viral particles (nominal dose) and at least 90 subjects per one intramuscular injection of rAd26-S at (10±0.5) 1*10^11 viral particles with a 4-week interval on study days 1 and 29, respectively.

Duration of the subject participation in the study will be 6 months (180±10 days) from the day of administration of the first dose of AZD1222 vaccine. 10 visits are scheduled for each subject, 8 of them being obligatory personal visits to the study site.

Safety will be assessed for the duration of the study as follows:

* Solicited adverse events (AEs) (local and systemic) will be assessed for 7 days following each vaccination (ie, on days 1-7 after the first vaccination and on study days 29-35 to account for AEs after second vaccination) at the study visits and based on the results of Subject Diary review.
* Unsolicited AEs will be recorded within 29 days after administration of each dose of AZD1222/rAd26-S vaccine (i.e. on days 1-29 and on days 29 to 57).
* Serious adverse events (SAEs) will be recorded from signing of the informed consent form through Day 180
* Adverse events of special interest (AESI) will be documented from the first vaccination until day 180.

Immunogenicity will also be assessed throughout the study and include serological assay of levels of antibodies specific for Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) antigen as well as level of seroconversion, tests for neutralising antibodies.

At least 100 subjects are expected to receive at least one dose of the study product in 1 study site on the territory of Republic Azerbaijan.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are:

   1. Overtly healthy as determined by medical examination, or
   2. Medically stable such that, according to the judgment of the investigator, hospitalisation within the study period is not anticipated and the participant appears likely to be able to remain in follow-up through the end of protocol-specified follow up.

   (A stable medical condition is defined as disease not requiring significant change in therapy or hospitalisation for worsening disease during the 3 months prior to enrolment.)
2. Able to understand and comply with study requirements/procedures based on the assessment of the investigator.
3. Female participants

   1. Women of childbearing potential must:

      * Have a negative pregnancy test on the day of screening and Day 1.
      * Use of a highly effective form of birth control for at least 28 days prior to Day 1 and agree to continue using one highly effective form of birth control through 60 days following administration of the second dose of study vaccine. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1 % per year when used consistently and correctly (see the table below). Periodic abstinence, the rhythm method, and withdrawal are NOT acceptable methods of contraception.
   2. Women are considered of childbearing potential unless they meet either of the following criteria:

      * Surgically sterilized (including bilateral tubal ligation, bilateral oophorectomy or hysterectomy) or
      * Postmenopausal
      * For women aged < 50 years old, postmenopause is defined as having both:

        * A history ≥ 12 months amenorrhea prior to the first dosing, without an alternative cause, following cessation of exogenous sex hormone treatment and
        * A follicle-stimulating hormone level in post-menopausal range. (Until follicle-stimulating hormone is documented to be within menopausal range, the participant is to be considered of childbearing potential.)
      * For women aged ≥ 50 years old, postmenopausal is defined as having a history of ≥ 12 months amenorrhea prior to first dosing, without an alternative cause, following cessation of exogenous sex hormone treatment.
4. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Known past confirmed SARS-CoV-2 infection less than 6 month prior to screening (the date of diagnosis must be confirmed by an official document).
2. Positive SARS-CoV-2 Reverse transcriptase polymerase chain reaction (RT-PCR) test at screening.
3. Significant infection or other illness including fever > 37.8 °C on the day prior to or day of vaccination.
4. Thrombocytopenia of grade ≥ 2 (i.e., <100,000/ mm3)
5. Clinically significant neutropenia (as determined by the investigator).
6. Clinically significant anemia (as determined by the investigator).
7. Any confirmed or suspected immunosuppressive or immunodeficient condition including infection caused by human immunodeficiency virus (HIV); asplenia; recurring and severe infections and administration of chronic immunosuppressive drugs within previous 6 months ( ≥ 20 mg/day of prednisone or another steroid at an equivalent dose used daily or every other day for ≥ 15 days within the 30-day period preceding immunization) except for topical/inhalation steroids or short-term oral steroids (courses ≤14 days).

   1. Note: enrollment of HIV-positive subjects with CD4 levels > 500 cells/mL3 ≥12 months receiving stable antiretroviral therapy for HIV therapy is allowed.
   2. Note: topical use of tacrolimus is permitted unless it was used within 14 days prior to enrollment.
8. History of allergic reactions to any of the product ingredients.
9. History of anaphylaxis or angioedema.
10. Current diagnosis of a malignant neoplasm and therapy thereof (except for basal-cell skin carcinoma or cervical cancer in situ).
11. History of serious mental conditions which are expected to impair participation in this study.
12. Bleeding disorders (e.g. coagulation factor deficiency, coagulopathy or impaired platelet disorders) or history of relevant hemorrhages or subcutaneous bruises after intramuscular injections or vein punctures.
13. Suspected alcohol or psychoactive drug addiction or a known current addiction.
14. History of Guillain-Barre syndrome or other demyelinating conditions.
15. Any other relevant diseases, disorders or findings which may significantly increase the risk due to participation in this study, restrict the subject's participation in it or impair interpretation of the study data.

    (Note: upon assessment of the subject for exclusion criterion No. 13, adverse events of special interest should be considered which are outlined in appendix F of the study protocol as these adverse events of special interest, particularly with no treatment or control, may pose a risk for the subject's safety. Restrict his/her participation in the study or impair interpretation of the study data. The investigator should be aware of the list of conditions given in Appendix E of the study protocol and take it into account. If any of these conditions are found in the subject, the Investigator will be asked to use his/her clinical judgement to decide on the subject's eligibility for the study. If a subject with conditions outlined in Appendix E of the study protocol is enrolled into the study, the Investigator will be asked to document the final justification for the enrollment in the site's medical document.)
16. Severe and/or uncontrollable cardiovascular diseases, respiratory diseases, gastrointestinal disorders, hepatic, renal, endocrine and nervous system diseases (mild/moderate adequately controlled co-morbidities are acceptable).
17. Prior splenectomy.
18. History of cerebral venous sinus thrombosis or experienced major venous and/or arterial thrombosis.
19. Any vaccines (authorized or experimental) other than the investigational ones within 30 days prior to and after each vaccination.
20. Previous or scheduled investigational or authorized vaccines or a product which may affect the interpretation of the study data (e.g. adenoviral vector-based vaccines, any coronavirus vaccines).
21. Administration of immunoglobulins and/or any blood components within 3 months prior to scheduled administration of the study vaccine.
22. Ongoing use of anticoagulants, e.g. coumarin and related ones (i.e. warfarin) or novel oral anticoagulants (e.g. apixaban, rivaroxaban, dabigatran and edoxaban).
23. Participation in studies of medicinal products for prevention of COVID-19 throughout the study.
24. Participation in planning and/or performance of this study (applicable to both Sponsor's personnel and/or study site personnel).
25. According to the Investigator, an individual should not participate in the study if the probability of compliance with study procedures, restrictions and requirements is low.
26. Previous participation in this study (undergoing screening and study inclusion procedures).
27. Female subjects only: current pregnancy (verified by positive pregnancy test) or breastfeeding.
28. Unwilling to refrain from blood donation during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Antibody seroconversion rate to SARS CoV-2 Spike protein 29 days after the second vaccination. | Day 57
  Antibody seroconversion rate (≥4-fold increase from baseline) to SARS CoV-2 Spike protein 29 days after the second vaccination.

SECONDARY OUTCOMES:
Incidence of local and systemic solicited Adverse Events (AEs) for 7 days post each dose | from Day 1 to Day 8 and From Day 29 to Day 36
  Number of Participants Reporting local (Pain at the site of injection, Erythema/hyperemia at the site of injection, Tenderness, Induration/swelling at the site of injection) and systemic (Fever > 37.8°C, Chills, Muscle pains, Fatigue, Headache, Malaise, Nausea, Vomiting) Solicited Adverse Events for 7 days following each vaccination (Day 1 through Day 7 for first vaccination and Day 29 through Day 35 for second vaccination).
Incidence of unsolicited AEs, serious adverse events (SAEs) and AEs of special interest | up to day 29, up to day 57
  Number of Participants Reporting unsolicited AEs, SAEs and AESIs through 29 days post each vaccination (i.e. up to day 29 after the first vaccination and day 57 after second vaccination).
Antibody seroconversion rate to SARS CoV-2 Spike protein 29 days after the first vaccination. | day 29
  The proportion of participants who have a post treatment seroresponse (defined as: ≥ 4 fold rise in titres from Day 1 baseline value) to the SARS CoV-2 Spike protein 29 days post first vaccination.
Antibody seroconversion rate against receptor-binding domain antigen 29 days after each vaccination. | day 29, 57
  The proportion of participants with post treatment seroresponse (defined as: ≥ 4-fold rise in titres from Day 1 baseline value) to receptor-binding domain antigen 29 days post each vaccination.
Change from baseline Geometric mean titre (GMT) values for evaluation of immunogenicity for Spike protein and receptor-binding receptor domain antigens | Day 1, 15, 29, 57, 180
  Сhange from baseline GMT values for evaluation of immunogenicity for Spike protein and receptor-binding receptor domain antigens at day 15, 29, 57, 180.
Change from baseline Geometric mean fold rise (GMFR) values for evaluation of immunogenicity for Spike protein and receptor-binding receptor domain antigens | Day 1, 15, 29, 57, 180
  Сhange from baseline GMFR values for evaluation of immunogenicity for Spike protein and receptor-binding receptor domain antigens at Day 15, 29, 57, 180.
Antibody seroconversion rate of neutralizing antibodies to SARS-CoV-2 antigen - 29 days after each vaccination | day 29, 57
  The proportion of participants with post treatment seroresponse (defined as: ≥ 4-fold rise in titres day from Day 1 baseline value to 29 days post each vaccination - Day 29 and Day 57), as measured by SARS-CoV-2 neutralising antibodies
Change from baseline GMT values for assessment of immunogenicity based of neutralizing antibodies to SARS-CoV-2 | Day 1, 15, 29, 57, 180
  Сhange from baseline GMT values for assessment of immunogenicity based of neutralizing antibodies to SARS-CoV-2 at Day 15, 29, 57, 180.
Change from baseline GMFR values for assessment of immunogenicity based of neutralizing antibodies to SARS-CoV-2 | Day 1, 15, 29, 57, 180
  Сhange from baseline GMFR values for assessment of immunogenicity based of neutralizing antibodies to SARS-CoV-2 at Day 15, 29, 57, 180.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — Chief Medical Officer, R-Pharm
Locations (1):
- Public legal entity "Baku Health Center", Baku, Azerbaijan